CLINICAL TRIAL: NCT02279784
Title: Drug Eluting Balloon in peripherAl inTErvention for Below-The-Knee Arteries With Freeway and Lutonix
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Leonardo Bolognese, MD, MD, Ospedale San Donato
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Arezzo013
Record Dates: First submitted 2014-10-28; First posted 2014-10-31 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Freeway (Experimental): angioplasty with Freeway drug-eluting balloon
  Interventions: Device: Freeway PTA
- Lutonix (Experimental): angioplasty with Lutonix drug-eluting balloon
  Interventions: Device: Lutonix PTA

INTERVENTIONS:
Device: Freeway PTA — angioplasty with Freeway drug-eluting balloon
  Arms: Freeway
Device: Lutonix PTA — angioplasty with Lutonix drug-eluting balloon
  Arms: Lutonix

SUMMARY:
The aim of this study is to compare in patients with critical limb ischemia the efficacy of angioplasty with different paclitaxel-eluting balloon devices for below-the-knee lesions in terms of restenosis.

DETAILED DESCRIPTION:
Two devices will be evaluated: the Lutonix and the Freeway paclitaxel eluting balloons. A post-hoc analysis will compare the results with the historical data from DEBATE-BTK (NCT01558505).

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* angiographic stenosis>50% or occlusion of one below-knee vessel

Exclusion Criteria:

* allergy to Paclitaxel
* contraindication for combined antiplatelet treatment
* life expectancy <1 year
* hypersensitivity or contraindication to one of the study drugs
* lack of consent
* need for amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
number of events of angiographic binary restenosis | 12 months
  number of events of angiographic binary restenosis

SECONDARY OUTCOMES:
number of events of target lesion revascularization | 12 months
  number of events of target lesion revascularization
number of events of death | 12 months
  number of events of death
frequency of major amputation | 12 months
  frequency of major amputation

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Department, Ospedale S.Donato, Arezzo, AR, Italy